CLINICAL TRIAL: NCT03644199
Title: Factors Responsible for the Development of Diabetes in Adults With Cystic Fibrosis
Brief Title: Development of Diabetes in Adults With Cystic Fibrosis (CF)
Acronym: CF-DIABETES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 11-NW-0552
Record Dates: First submitted 2016-05-10; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Cystic Fibrosis
Keywords: Gastric emptying; Cystic Fibrosis related diabetes; Incretins
MeSH Terms: conditions — Cystic Fibrosis | interventions — Glucose Tolerance Test

ARMS (2):
- OGTT test (Other): Comparison of responses to a OGTT between CF subjects and health control subjects
  Interventions: Other: Oral Glucose Tolerance Test (OGTT) assessment arm
- Mixed meal (Other): Comparison of responses to a mixed meal through the day between CF subjects and health control subjects
  Interventions: Other: Mixed meal test evaluation test arm

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) assessment arm — Hormonal and motility responses to a standard OGTT evaluation arm
  Arms: OGTT test
Other: Mixed meal test evaluation test arm — Evaluate the hormonal and motility responses to a standard mixed meal test through the day
  Arms: Mixed meal

SUMMARY:
This is a crossover study to determine the possible factors that might be related to the development of diabetes in CF and examines the relationship between pancreatic fatigue if any, and the development of diabetes. In addition hormones affecting the release of insulin and stomach motility will be studied to determine if there is a variation in response to solid and liquid meals and if this variation increases as fatigue progresses.

DETAILED DESCRIPTION:
The main purpose of this study is to look at possible additional factors that might be related to the development of Cystic Fibrosis Related Diabetes (CFRD), that in itself is a unique entity and to identify an appropriate test to diagnose CFRD. There is well demonstrated evidence of delayed insulin release and peak in individuals with CF, the cause of which is not fully explained.

With a view to determine the cause of this phenomenon the aims of this study are:

1. To determine whether pancreatic fatigue contributes to this delayed insulin release and peak that is seen in patients with cystic fibrosis.
2. Should a glucose tolerance test be done at a later time in the day, as against first thing in the morning as is the current accepted standard?
3. To determine if gastric emptying has a role to play in the development of CFRD?
4. To study the hormone release response to a glucose challenge and the patterns of change through the day.
5. To study the relationship of these hormones to gastric emptying and the development of diabetes.

ELIGIBILITY:
In order to participate in the study, the CF group must meet all the following inclusion criteria

1. Male or female with a confirmed diagnosis of cystic fibrosis defined by

   1. Clinical features consistent with a diagnosis of CF AND
   2. Sweat chloride ≥60mmol/L by pilocarpine ionotophoresis; OR
   3. Genotypic confirmation of CFTR mutation
2. Aged 18 - 50 years
3. Out-patients from the regional adult unit in Liverpool
4. Currently not known to be diabetic or on insulin
5. Clinically stable over the preceding 4 weeks i.e. no indication for iv antibiotics, steroids or hospital admissions
6. Hemoglobin value >10g/dl

The inclusion criteria for the normal population group is as follows:

1. Male or female with NO confirmed diagnosis of cystic fibrosis
2. Aged 18 - 50 years
3. Currently not known to be diabetic or on insulin
4. Clinically stable over the preceding 4 weeks i.e. no indication for iv antibiotics, steroids or hospital admissions
5. Hemoglobin value >10g/dl

In order to participate subjects must not meet any of the following exclusion criteria

1. Patients with known diabetes or on glucose lowering medications (insulin, oral agents)
2. On-going acute illness
3. Those on long-term oral steroids
4. Pregnant women
5. Those on immunosuppressive treatment
6. History of, or planned organ transplant
7. Clinically significant abnormal findings on haematology or clinical chemistry
8. Subjects with documented or suspected, clinically significant, alcohol or drug abuse. The determination of clinical significance will be determined by the investigator.
9. Current malignant disease
10. Any serious or active medical or psychiatric illness, which in eth opinion of the investigator, would interfere with subject treatment, assessment, or compliance with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03-30 (Estimated); Primary Completion 2013-07-30 (Estimated); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Glucose levels | 4 hours
  Glucose sensitivity test

SECONDARY OUTCOMES:
Insulin responses | 4 hours
  Insulin resistance test
GLP1 and GIP responses | 4 hours
  GLP1 and GIP tests
Evaluation of gastric emptying | 8 hours
  Gastric flow measurement

CONTACTS AND LOCATIONS:
Overall Officials: Dilip Nazareth, MD, Principal Investigator — Liverpool Heart & Chest Hospital
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided